CLINICAL TRIAL: NCT03757052
Title: Safety, Validity and Efficiency of a Direct Graded Oral Challenge With Amoxicillin for the Evaluation of Penicillin Allergy in Adults
Brief Title: Amoxicillin Challenge for Penicillin Allergy Diagnosis
Acronym: Pen-VIE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-4379
Record Dates: First submitted 2018-11-22; First posted 2018-11-28 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Penicillin Allergy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Skin testing and Graded Oral Challenge (Experimental): Penicillin skin testing as described in the intervention section, followed by amoxicillin graded oral challenge as described in the intervention section
  Interventions: Diagnostic Test: Penicillin Skin Testing

INTERVENTIONS:
Diagnostic Test: Penicillin Skin Testing — Skin test protocol: prick skin tests (penicilloyl-polylysine 0.000012 mol/0.05 mL, penicillin G 10,000 U/mL, penoate 10,000 U/mL, ampicillin 100 mg/mL, amoxicillin 71 mg/mL, histamine/positive control, diluent/negative control), then intradermal skin tests (penicilloyl-polylysine 0.000012 mol/0.05 mL, penicillin G 10,000 U/mL, penoate 10,000 U/mL, ampicillin 1 mg/mL, diluent/negative control), administered as an intradermal injection of a standardized volume of 0.02 mL. Graded oral challenge with amoxicillin : a first dose of 50 mg of amoxicillin; 20-minute observation period; in the absence of any objective symptom of an allergic reaction, a second dose of amoxicillin of 450 mg; final observation period of 60 minutes, under nurse and medical supervision.
  Other Names: Amoxicillin Graded Oral Challenge

SUMMARY:
False diagnosis of penicillin allergy are frequently reported, and have been proven detrimental to patients. Current guidelines for the assessment of drug allergies recommend that penicillin allergy be evaluated first with prick and intradermal skin tests, and then completed with a graded oral challenge, spread over at least two doses. However, it has been shown that these skin tests, in addition to consuming resources and time, are of limited, or even doubtful validity, given the poor predictive values that have been reported in the modern penicillins era. It now seems unreasonable to continue their use without addressing other, more efficient diagnostic stategies. Several groups have now demonstrated the safety, validity, and efficiency of a direct, two-step amoxicillin oral challenge (starting with 10% of the standard therapeutic dose, followed by 90 % of the dose), without prior skin tests, first for any type of reaction in the pediatric population, then for any non-immediate reaction in the adult population. The objective of this study is to demonstrate the safety, efficiency, and validity of direct, two-step graded oral challenge with amoxicillin for the evaluation of any reported penicillin allergy in the adult population, excluding high-risk patients (documented anaphylaxis to a penicillin in the last 5 years). Skin tests will first be performed according to the protocol currently in use at the CHUL, then consented patients will proceed with the graded oral challenge still according to the protocol currently in use at the CHUL, but regardless of the skin tests results. The results of the two tests will be compared to determine the safety, efficiency and validity of proceeding directly to the graded oral challenge.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older at the time of the test
* Being referred by a health professional for the evaluation of any allergic reaction to a penicillin, including natural penicillins, anti-staphylococcal penicillins, aminopenicillins, penicillins combined with a beta-lactamase inhibitor, and carboxypenicillins ; or an antibiotic of the beta-lactam family, whose assessment requires testing for penicillins, according to the treating allergist

Exclusion Criteria:

* Pregnancy
* Poorly controlled asthma, chronic lung disease or heart disease
* Failure to stop beta-blockers prior to the test
* Occurrence of the reaction in the 4 weeks preceding the test (possibility of false negatives)
* History of severe delayed hypersensitivity reaction, reaction requiring hospitalization of more than 24 hours, or bullous, pustular, exfoliative or mucosal reaction (excluding angioedema)
* Recent anaphylaxis (<5 years), defined as concomitant involvement of at least two systems (respiratory, digestive, mucocutaneous or cardiovascular) within one hour of administration of the drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Type 1 Hypersensitivity Reaction | 60 minutes
  The primary outcome is the occurrence of immediate hypersensitivity symptoms, occuring during the test period, which is up to 60 minutes after the last dose of amoxicillin.

SECONDARY OUTCOMES:
Skin Tests Results | 60 minutes
  Concordance of Skin Tests Results with Oral Challenge Results
Severity of immediate hypersensitivity symptoms | 60 minutes
  Mild, moderate and severe
Delayed hypersensitivity symptoms | 14 days
  Occurrence of delayed hypersensitivity symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Drolet, MD FRCPC, Principal Investigator — CHU de Quebec-Universite Laval
Locations (1):
- CHU de Quebec, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided